CLINICAL TRIAL: NCT05847530
Title: Pilot Evaluation of the Cynosure Potenza™ System for Treatment of Cosmetic Dermatologic Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-PL01-2022
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Wrinkles; Scars; Stretch Marks; Pigmentation; Skin Laxity
MeSH Terms: conditions — Cicatrix; Striae Distensae; Cutis Laxa

STUDY DESIGN:
Intervention Model Description: Randomization is not requires, as the group to which a subject is assigned to will be at the discretion of the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Experimental): This group is Potenza treatments only.
  Interventions: Device: Potenza
- Group B (Experimental): This group is Potenza and Icon treatments.
  Interventions: Device: Potenza; Device: Icon

INTERVENTIONS:
Device: Potenza — Subjects will receive 1-4 treatments at approximately 1 month intervals, but other intervals from 2 to 12 weeks may take place at the PI's discretion. At the discretion of the PI, additional follow-up visits may take place to observe the time course of skin reactions after treatment and/or to assess if the skin condition continues to improve beyond 3 months after treatment.
Device: Icon — Subjects will receive 1-4 treatments at approximately 1 month intervals, but other intervals from 2 to 12 weeks may take place at the PI's discretion. At the discretion of the PI, additional follow-up visits may take place to observe the time course of skin reactions after treatment and/or to assess if the skin condition continues to improve beyond 3 months after treatment.
  Arms: Group B

SUMMARY:
The primary objective of this pilot study is exploratory investigation evaluating the Potenza microneedle fractional radiofrequency (RF) device and may be used in combination with the Icon intense pulsed light (IPL) device.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female 18 years of age or older.
* Presence of unwanted dermatologic condition suitable for treatment such as facial and/or neck wrinkles, skin laxity of face, neck or body, scars, acne scars or striae, or Vascular and/or pigment dyschromia
* Ability to read, understand, and sign the Informed Consent Form
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated and/or weight loss through the follow-up period.
* Willing and able to comply with all study participation requirements including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using (or willing to use) medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* Presence of an active systemic or local skin disease or condition that may affect wound healing or interfere with participation.
* History of keloids or poor wound healing
* Taking medication which is known to increase sensitivity to sunlight
* Has a seizure disorders triggered by light
* Cancer, malignant disease, skin pathology, condition or allergic reactions that could interfere with evaluation or with the use of typical ancillary medical treatments or care used before, during or after treatments
* History of collagen, vascular or immunosuppressive or deficiency disorders
* History of coagulative disorder or use of anticoagulant drugs within 2 weeks of study treatment
* Use of steroids within 2 weeks of study treatments
* Use of Accutane (isotretinoin) in the past 12 months
* Previous surgical or cosmetic procedure to the target area in the last 6 to 12 months that could interfere with the treatment procedure and affect treatment outcome
* Has an implanted pacemaker or defibrillator, metal pins or prosthetic joints
* Allergic reaction to gold metal
* Receiving or have received gold therapy
* Photo-sensitive skin
* Psycho-neurotic condition including alcohol or drug abuse
* Unwilling or unable to adhere to all study requirements for treatment and follow-up
* Has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Grading of Skin Aging and Photodamage | 90 days post last treatment
  At the 90 day follow up, subjects will be graded on a scale of 0-4 (0 being none and 4 being severe) for the presence of skin aging and photodamage. The # of subjects with improvement will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Clinic, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No